CLINICAL TRIAL: NCT02618863
Title: The Cricoid Force Necessary to Occlude the Esophageal Entrance: Is There a Gender Difference?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, Dr.AHED ZEIDAN, Procare Riaya Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRH7
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: ASPIRATION

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 , cricoid pressure (Active Comparator): 30 male
  Interventions: Device: Cricoid pressure
- 2,cricoid pressure (Active Comparator): 30 female
  Interventions: Device: Cricoid pressure

INTERVENTIONS:
Device: Cricoid pressure — Applying cricoid pressure and testing its effectiveness using gastric tube . in addition , by using the cricometer , the CP 50 is defined and compared in both gender

SUMMARY:
the investigators have observed that women may require less CF than men to occlude the esophageal entrance, and that the routine use of 30 N in women may actually increase the incidence of airway-related problems. The objective of the current investigation was to test this hypothesis. In this study, real-time visual and dynamic means were used to assess the effectiveness of different forces applied to the cricoid cartilage in occluding the esophageal entrance in men and women. The patency of the esophageal entrance was directly visualized using the Glidescope Video Laryngoscope in anesthetized and paralyzed patients with and without CP. Evidence of closure of the esophageal lumen was confirmed by the inability to introduce a gastric tube (GT) into the esophagus under direct vision. New method , using Cricometer , was used to measure the applied force .

DETAILED DESCRIPTION:
60 (30 men; ages 18 - 50 yr; body mass index < 28 kg/m2 physical status 1, 2 patients were recruited for the study. These patients were to undergo general anesthesia with tracheal intubation. starting force was 20 N in both sex. These forces were standardized by reproducing a new device : cricometer. The sequence of the applied forces was done by using the up and down method in both sex. After preoxygenation, anesthetic induction, muscular relaxation and mask ventilation, the study commenced. Direct laryngoscopy using the Glidescope video laryngoscope was performed and the view of the glottis and the esophageal entrance was video recorded with each CF. 2 attempts to insert a lubricated gastric tube (GT; size 20 F, 12 F) were carried out by a "blinded" operator in each patient. A successful insertion of the GT indicated a patent esophagus. When this occurred while CP was applied, it indicated ineffective CP. An unsuccessful insertion of the GT while CP was applied indicated a non-patent esophagus (effective CP). The position of the esophageal entrance relative to the glottis during CP was assessed from the video recordings.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 2
* Easy Identification cricoid cartilage
* No contre indication to CP

Exclusion Criteria:

* obese patients
* ASA2 & ASA3
* contre indication to CP

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Necessary force of CP to occlude the esophagus in female versus male . an up and down method will define the CP 50 in each gender . A comparison between CP50 in both sex will define exactly our outcome : Is there a gender difference . | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: kamal abdulkhaleq, MD, Study Director — Procare Riaya Hospital
Locations (1):
- Procare Riaya Hospital, Khobar, Estern, Saudi Arabia

REFERENCES:
- [Derived] Zeidan AM, Salem MR, Bamadhaj M, Mazoit JX, Sadek H, Houjairy H, Abdulkhaleq K, Bamadhaj N. The Cricoid Force Necessary to Occlude the Esophageal Entrance: Is There a Gender Difference? Anesth Analg. 2017 Apr;124(4):1168-1173. doi: 10.1213/ANE.0000000000001631. PMID 28079588